CLINICAL TRIAL: NCT00456157
Title: A Phase 1, Double-Blind, Randomized, Single Dose Escalation Safety Study of Intra-articular Osteogenic Protein-1 OP-1 in Subjects With Osteoarthritis of the Knee
Brief Title: A Phase 1, Double-Blind, Randomized, Single Dose Escalation Safety Study of Intra-articular OP-1 in Subjects With Osteoarthritis of the Knee
Acronym: Knee OA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stryker Biotech (Industry)
Responsible Party: Gina Smith, Stryker Biotech
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 06-OA-001
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Osteophytes; Knee; Intra-articular; OP-1
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Osteophyte

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Intra-articular Injection of OP-1 to affected knee

SUMMARY:
The purpose of this research study is to investigate the safety and tolerability of OP-1 when it is injected into the knee joint of patients who have osteoarthritis on the knee.

DETAILED DESCRIPTION:
Subjects with OA will be recruited and informed consent obtained. During a screening period lasting 1 to 28 days, subjects will undergo medical and arthritis history, physical examination, collection of concomitant medications, KOOS (which contains the WOMAC questionnaire), SF-36 and global 100 mm VAS assessments, have samples obtained for urinalysis, hematology, chemistry, immunology and serum and plasma for future biomarker testing, ECG, bilateral knee x-rays and MRI of the index knee at selected sites. Subjects who meet all of the inclusion criteria and none of the exclusion criteria will be randomized into the first cohort of 8 subjects to receive either 1.0 mL lactose (placebo) (2 subjects) or 1.0 mL OP-1 (6 subjects) intraarticularly using ultrasound or fluoroscopy guidance in an outpatient setting on day 1. Each cohort will consist of 8 treated patients, with treatment allocation in a 3:1 active-to-lactose (placebo) ratio. After an observation period of at least one hour, subjects will be released and contacted via telephone on Day 2 to query for AEs and concomitant medications. Additional follow-up visits will be done on days 7, 14, 28, 56, 84 and 168 (weeks 1, 2, 4, 8, 12 and 24) and safety and efficacy parameters evaluated according to the Schedule of Events. When a minimum of 4 weeks have elapsed since the last patient of the current cohort has been treated, all safety data will be collected and reviewed by the Principal Investigators and the Sponsor. The safety review will be conducted to ensure the demonstrated safety profile of OP-1 is acceptable for the treated patients. Only after the current dose level has been judged to be safe will dose escalation to the next dosing cohort occur.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory subjects with OA of the knee with symptoms for at least 6 months and pain on the majority of days in the last 30 days. Symptoms must include knee joint pain, and may include crepitus, swelling and/or effusion of the knee. In subjects with bilateral knee OA, the more symptomatic knee is the index knee. Subjects may be taking NSAIDs, analgesics and/or undergoing physical therapy.
* Age > 40 years
* Radiographic evidence on posteroanterior (PA) and lateral standing, flexed x-rays of at least one osteophyte.
* Subjects must be willing to abstain from other intraarticular treatments of the knee or any surgery for 12 weeks on study.
* Ability to comply with the study and give informed consent.
* Subjects must be willing to abstain from NSAIDs or analgesic medications (except for acetaminophen) for 48 hours prior to assessments, at screening, day 1 and week 4, 8, 12, and 24 visits.

Exclusion Criteria:

* Concurrent medical or arthritic conditions which could interfere with evaluation of the index knee joint including fibromyalgia.
* Subject has received arthroscopic or open surgery to the index joint within 6 months of study start
* The presence of surgical hardware or other foreign body in the index joint
* Corticosteroid, hyaluronic acid or other intraarticular injection within 3 months of study start
* Use of chondroitin and/or glucosamine within 4 weeks prior to study start
* History of Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, lymphoma, arthritis associated with inflammatory bowel disease, sarcoidosis or amyloidosis
* Clinical signs and symptoms of active knee infection or crystal disease
* Clinically significant cardiac disease, consult study Medical Monitor
* Have an increased predisposition for the development of infections
* History of malignancy, with the exception of resected basal cell carcinoma, squamous cell carcinoma of the skin, or resected cervical atypia or carcinoma in situ.
* More significant pain from the back or the hip than the knee
* Skin breakdown at the knee where the injection would take place
* Planned knee replacement during the study period
* For subjects undergoing MRI, the presence of contraindications to having an MRI at the specific imaging facility.
* For subjects undergoing MRI, an estimated Glomerular Filtration Rate (eGFR) of <45 mL/min calculated using the Cockcroft-Gault estimate for eGFR as follows:

eGFR = (140-age [yrs]) X weight [kg] / serum creatinine [mg/dL] X 72 (X 0.85 for women)

* For subjects undergoing MRI, known allergy to gadolinium contrast material
* Has known or clinically suspected infection with human immunodeficiency virus (HIV), hepatitis C or B viruses
* Has participated within 30 days or will participate concurrently in another investigational drug or vaccine study
* Has a history of drug or alcohol dependence in the past 3 years
* Known sensitivity to lidocaine or OP-1
* Female with reproductive capability
* Has other serious, non-malignant, significant, acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.
* Prior use of a bone morphogenetic protein.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2007-03; Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Determine safety and tolerability as well as dose limiting toxicity (DLT) and maximal tolerated dose (MTD) of intraarticular OP-1

SECONDARY OUTCOMES:
Determine the proportion of patients with 20%, 50%, and 70% improvement in the Western Ontario and McMaster (WOMAC) pain, and function subscales at 4, 8, 12, and 24 weeks.
Determine the change from baseline to 4, 8, 12, and 24 weeks in the pain, other symptoms, function in daily living, function in sports and recreation and knee related quality of life subscales of the Knee and Osteoarthritis Outcome Score (KOOS) survey.
Determine the change from baseline to 4, 8, 12, and 24 weeks in the patient's global assessment and disease status and physician's global assessment and disease status using the 100-mm visual-analogue scale (VAS).
Quality of life measured by the Short Form (SF)-36 at baseline and 4, 8,12 and 24 weeks
Amount of rescue medications required at 4, 8, 12 and 24 weeks
Knee cartilege and surrounding saft tissue changes by magnetic resonance imaging (MRI) of the index knee and proteoglycan content by delayed gadolinium enhanced MRI of cartilage (dGEMRIC)
Analysis of efficacy data using the Outcome Measures in Arthritis Clinical Trials -Osteoarthritis Research Society (OMERACT-OARSI) Responder Index
Blood levels of OP-1

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - University of orth Carolina School of Medicine, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Hunter DJ, Pike MC, Jonas BL, Kissin E, Krop J, McAlindon T. Phase 1 safety and tolerability study of BMP-7 in symptomatic knee osteoarthritis. BMC Musculoskelet Disord. 2010 Oct 10;11:232. doi: 10.1186/1471-2474-11-232. PMID 20932341